CLINICAL TRIAL: NCT03426293
Title: MANCO: Measuring the ACT During Non-cardiac Arterial Procedures.
Brief Title: Measuring the ACT During Non-cardiac Arterial Procedures.
Acronym: MANCO
Status: Completed | Type: Observational
Sponsor: Dijklander Ziekenhuis (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Arno Wiersema, Principal Investigator, Dijklander Ziekenhuis
Other Study IDs: M016-045
Record Dates: First submitted 2018-01-27; First posted 2018-02-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Arterial Disease; Surgery; PTA; Peripheral Arterial Disease
Keywords: heparin;ACT;non-cardiac vascular;peri-procedural
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arterial procedure and ACT measurement: All patients undergoing an open or endovascular arterial procedure in which heparin is used peri-procedurally and the ACT is measured to determine effect of heparin
  Interventions: Other: Measuring the ACT to determine effect of heparin

INTERVENTIONS:
Other: Measuring the ACT to determine effect of heparin — Measuring the ACT to determine effect of heparin during non-cardiac arterial procedures

SUMMARY:
Aim of the MANCO study is to establish for once and for all that monitoring the effect of heparin during NCVI (Non-Cardiac Vascular Interventions) is essential to ensure the individual patient of safe and tailor-made anticoagulation. Not measuring the effect of the administered heparin exposes the patient to unnecessary risks of thrombo-embolic and bleeding complications. First aim of the MANCO study is to prove that the standardized bolus of 5000 IU of heparin, used by 90% of vascular specialists in Europe, results in inadequate anticoagulation in more than 80% of patients. These measurements will be performed using the Hemostasis Management System by Medtronic.

DETAILED DESCRIPTION:
Heparin is used worldwide by all vascular surgeons and interventional radiologists (IR) during non-cardiac vascular interventions (NCVI), both open and endovascular. Heparin is used to reduce or prevent arterial thrombo-embolic complications (ATEC). Heparin reduces the clotting of blood and thereby coagulation. This also explains the negative side-effect of using heparin: its use can lead to bleeding-complications, possibly causing the need for blood tranfusions, more hematomas necessitating re-interventions and increasing the risk of infections.

Since the 1970's it is well known that heparin has a non-linear dose response curve and also a non-linear elimination curve in the individual patient.

Despite this fact, more than 95% of all vascular surgeons and IR use a standardized bolus of 5000 IU in every patient. Multiple studies have demonstrated that up to 70% of patients is not adequately anticoagulated during NCVI using that bolus of 5000 IU.

During open or endovascular cardiac interventions the effect of heparin is always routinely measured using the activated clotting time (ACT).

Despite this knowledge the percentage of vascular surgeons and/or IR that measure the effect of heparin during NCVI routinely is astonishing low: 0-5%, in the US this percentage is probably higher (30%), possibly due to medico-legal reasons. Existing guidelines on NCVI depict different regimes on the use of heparin or do not mention this use at all.

The Hemostasis Management System (HMS, Medtronic) measures the ACT, but it also calculates a heparin dose response curve in the individual patient. This curve supplies the vascular surgeon or IR a tool to administer the exact amount of heparin needed to reach a desired ACT. Also the exact dose of protamine can be calculated to neutralize the effect of remaining circulating heparin in the individual patient. The use of the HMS in cardiac vascular procedures has to led to a reduced need for blood transfusions, less postoperative bleeding complications and a reduction of peri-procedural myocardial infarctions and other ATEC.

To determine if the HMS can be of equal high value during NCVI, a pilot study was performed at the VUMC, called Hepvasc. Results of this pilot (submitted) and other sparse results from literature, show that HMS can be used during NCVI. Furthermore, results indicated that the bolus of 5000 IU resulted in inadequate anticoagulation in 7 out of 18 included patients. This exposes those patients to a higher risk of ATEC.

As a result of this pilot, the MANCO study is designed with the HMS during NCVI. The MANCO study will evaluate the data of heparin management with the HMS in number of large vascular centers, starting in the Netherlands and after that in Europe. Measurements with the HMS will be used for the evaluation of the local heparin protocol by the individual vascular surgeon or IR. The MANCO study will be started permitting every center to apply their current heparin protocol. This includes the dosage of heparin and possible extra dosing of heparin to reach a desired ACT. The MANCO study is started as a prospective data registry and observational study of the ACT with an extensive case record form (CRF). Regular blood samples for ACT measurements will be done, so no extra invasive measurements are performed in the patient. Data will be collected according to all legal requirements and permission of local medical ethics committees is granted.

ELIGIBILITY:
Inclusion Criteria:

* All patients in participating centers undergoing Non-Cardiac Vascular (arterial) Intervention open or endovascular, older than 18 years

Exclusion Criteria:

* Patients with a known history of coagulation disorders or a EGFR lower than 30 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - All patients in participating centers undergoing NCVI, older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change of Activated Clotting Time | ACT measured before heparin, 5 minutes after and than at 30 minutes intervals. After a repeated dose of heparin again after 5 minutes and 30 minutes intervals
  Change of Activated Clotting Time, before and after administration of heparin

SECONDARY OUTCOMES:
Complications | 30 days or same admission, 6 weeks, 6 months and 12 months
  All complications as depicted in Suggested Standards for reports on arterial procedures and local complication registration. Vascular and non-vascular

CONTACTS AND LOCATIONS:
Overall Officials: Arno M Wiersema, MD, PhD, Principal Investigator — Dijklander Ziekenhuis
Locations (3):
- Netherlands (3):
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Westfriesgasthuis, Hoorn, North Holland
  - Isala klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
All ACT values can be obtained after trial with PI
Supporting Information: Study Protocol, SAP
Time Frame: after completion
Access Criteria: mail PI

REFERENCES:
- [Background] Wiersema AM, Watts C, Durran AC, Reijnen MM, van Delden OM, Moll FL, Vos JA. The Use of Heparin during Endovascular Peripheral Arterial Interventions: A Synopsis. Scientifica (Cairo). 2016;2016:1456298. doi: 10.1155/2016/1456298. Epub 2016 Apr 17. PMID 27190678
- [Background] Wiersema A, Jongkind V, Bruijninckx C, Reijnen M, Vos J, Van Delden O, Zeebregts C, Moll F. Prophylactic intraoperative antithrombotics in open infrainguinal arterial bypass surgery: a systematic review. J Cardiovasc Surg (Torino). 2015 Feb;56(1):127-43. Epub 2014 Mar 4. PMID 24594802
- [Background] Wiersema AM, Vos JA, Bruijninckx CMA, van Delden OM, Reijnen MMPJ, Vahl A, Zeebregts CJ, Moll FL. Periprocedural prophylactic antithrombotic strategies in interventional radiology: current practice in the Netherlands and comparison with the United kingdom. Cardiovasc Intervent Radiol. 2013 Dec;36(6):1477-1492. doi: 10.1007/s00270-013-0558-6. Epub 2013 Feb 13. PMID 23404518
- [Background] Wiersema AM, Jongkind V, Bruijninckx CM, Reijnen MM, Vos JA, van Delden OM, Zeebregts CJ, Moll FL; CAPPAStudy Group Consensus on Arterial PeriProcedural Anticoagulation. Prophylactic perioperative anti-thrombotics in open and endovascular abdominal aortic aneurysm (AAA) surgery: a systematic review. Eur J Vasc Endovasc Surg. 2012 Oct;44(4):359-67. doi: 10.1016/j.ejvs.2012.06.008. Epub 2012 Jul 24. PMID 22831869
- [Background] Finley A, Greenberg C. Review article: heparin sensitivity and resistance: management during cardiopulmonary bypass. Anesth Analg. 2013 Jun;116(6):1210-22. doi: 10.1213/ANE.0b013e31827e4e62. Epub 2013 Feb 13. PMID 23408671
- [Background] Mabry CD, Thompson BW, Read RC. Activated clotting time (ACT) monitoring of intraoperative heparinization in peripheral vascular surgery. Am J Surg. 1979 Dec;138(6):894-900. doi: 10.1016/0002-9610(79)90318-0. PMID 507308
- [Background] Goldhammer JE, Zimmerman D. Pro: Activated Clotting Time Should Be Monitored During Heparinization For Vascular Surgery. J Cardiothorac Vasc Anesth. 2018 Jun;32(3):1494-1496. doi: 10.1053/j.jvca.2017.04.047. Epub 2017 Apr 26. No abstract available. PMID 28943189
- [Background] Veerhoek D, Groepenhoff F, van der Sluijs MGJM, de Wever JWB, Blankensteijn JD, Vonk ABA, Boer C, Vermeulen CFW. Individual Differences in Heparin Sensitivity and Their Effect on Heparin Anticoagulation During Arterial Vascular Surgery. Eur J Vasc Endovasc Surg. 2017 Oct;54(4):534-541. doi: 10.1016/j.ejvs.2017.07.006. Epub 2017 Aug 9. PMID 28802634